CLINICAL TRIAL: NCT06162156
Title: The Effect of Back Massage After Cesarean on Pain, Anxiety, Sleep, Breastfeeding, Comfort, Uterine Involution and Physiological Parameters
Brief Title: Effects of Back Massage After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Esra Guler, PhD student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OÜ-HEM-EG-02
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Cesarean Section
Keywords: cesarean section; breastfeeding; sleep; anxiety; pain; comfort; uterine involution; back massage; physiological parameters
MeSH Terms: conditions — Breast Feeding; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: two groups with back massage experimental group and control group
Who Masked: Outcomes Assessor
Masking Description: Which group will be the intervention group and which group will be the control group will be determined by lottery. After the participant agrees to participate in the research, the person will draw envelopes from sealed envelopes by lottery and thus it will be determined which group he/she is in. Since the researcher and the mothers, who are massage practitioners, knew which group they were included in, the data collection phase of the study could not be blinded. Since the statistical analysis of the study will be performed by an independent statistician other than the researcher, the statistical analysis phase is blind. Therefore, the study is single blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- back massage group (Experimental): Volunteer women who meet the inclusion criteria after cesarean delivery will be selected by a random method, and verbal and written consent will be obtained from those included in the intervention group. Pre-test data twelve hours after cesarean delivery: 'Personal Information Form', 'Trait-Trait Anxiety Inventory', 'Postpartum Comfort Scale (PCS)', 'Bristol Breastfeeding Assessment Tool (BBAT)', 'Uterine Involution Evaluation Form ( UIEF)' 'Physiological Parameter Form (PPF)' and 'Visual Analog Scale (VAS)' will be filled in by the participants themselves using face-to-face interview technique in approximately twenty minutes. The intervention group will receive a twenty-minute back massage after the initial data is received. One hour after the massage, 'VAS' and 'PPF data will be filled in again. Post-test data twenty-four hours after the massage; 'Richard Campbell Sleep Scale', 'VAS, 'Trait-Trait Anxiety Inventory', 'PCS', 'BBAT, 'UIEF, 'PPF will be filled in again..
  Interventions: Other: Back massage
- control group (No Intervention): Volunteer women who meet the inclusion criteria after cesarean delivery will be selected by random method, and verbal and written consent of those included in the control group will be obtained. Pre-test data twelve hours after cesarean delivery: 'Personal Information Form', 'Trait-Trait Anxiety Inventory', 'Postpartum Comfort Scale (PCS)', 'Bristol Breastfeeding Assessment Tool (BBAT)', 'Uterine Involution Evaluation Form ( UIEF)' 'Physiological Parameter Form (PPF)' and 'Visual Analog Scale (VAS)' will be filled in by the participants themselves using face-to-face interview technique in approximately twenty minutes. The control group will not be massaged anywhere in the study. Thirteen hours after cesarean delivery, 'VAS' and 'PPF data will be filled in again. Posttest data twenty-four hours after cesarean delivery; 'Richard Campbell Sleep Scale', 'VAS, 'Trait-Trait Anxiety Inventory', 'PCS', 'BBAT, 'UIEF, 'PPF will be filled in again.

INTERVENTIONS:
Other: Back massage — For the intervention group, massage will be given to the participant's back area by the researcher for 20 minutes, 12 hours after the cesarean birth. Preliminary data forms will be filled out by the participant before the massage. One hour after the massage, 'Visual Analog Scala' and 'Physiological Parameter Form' data will be filled in again. The final data forms will be filled out by the participant 24 hours after the cesarean birth, that is, 12 hours after the back massage.
  Arms: back massage group

SUMMARY:
The aim of this study is to examine the effect of back massage application after cesarean section on women's pain, anxiety, sleep, breastfeeding, comfort, uterine involution process and physiological parameters. This research is a randomized controlled experimental type study with a pretest-posttest control group. In the research, after obtaining the necessary permissions and the ethics committee report, the application will be carried out to women who have given birth by cesarean section at the State Hospital and meet the criteria for inclusion in the study. Personal Information Form, Richard Campbell Sleep Scale, Trait-Trait Anxiety Inventory, Postpartum Comfort Scale, Bristol Breastfeeding Evaluation Tool, Visual Analog Scale for Pain, Uterine Involution Evaluation Form, Physiological Parameter Form will be used in the research.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of back massage after cesarean section on women's pain, anxiety, sleep, breastfeeding, comfort, uterine involution process and physiological parameters. This research is a randomized controlled experimental type study with a pretest-posttest control group. Personal Information Form, Richard Campbell Sleep Scale, Trait-Trait Anxiety Inventory, Postpartum Comfort Scale, Bristol Breastfeeding Evaluation Tool, Visual Analog Scale for Pain, Uterine Involution Evaluation Form, Physiological Parameter Form will be used in the research.

Collection of Data This research is a randomized controlled experimental type study with a pretest-posttest control group. The data of the research will be collected after the necessary institutional permission and ethics committee approval have been obtained. Data will be collected in three stages. Women who meet the inclusion criteria for the study will be informed about the method to be followed in the research. Those who want to participate in the research will read and sign the volunteer information form.

First Stage:

Women who apply to the selected hospital, meet the inclusion criteria and agree to participate in the study will be visited 12 hours after cesarean delivery, the women will be informed, verbal and written consent will be obtained from women who want to participate in the study, and pre-test data will be collected by the researcher. Before randomization to the intervention and control groups, the researcher will give general information to the mothers about the research at the 12th hour after cesarean section and their written informed consent will be obtained. The pre-test data of the research were collected face to face in an average of 20 minutes with the 'Personal Information Form', 'Trait-Trait Anxiety Inventory', 'Postpartum Comfort Scale', 'Bristol Breastfeeding Evaluation Tool', 'Uterus Involution Evaluation Form' and 'Physiological Parameter Form'. It will be filled in by the participants themselves using the interview technique. The height of the fundus section of the uterus, heart rate, body temperature, oxygen saturation, respiratory rate and blood pressure physiological parameters will be monitored by the researcher.

Second Stage:

'Visual Analog Scala' and 'Physiological Parameter Form' data will be filled in again by the researcher one hour after massage for the intervention group (13 hours after cesarean delivery), and for the control group 13 hours after cesarean delivery.

Third Stage:

Post-test data 24 hours after the intervention group was massaged by the researcher; 'Richard Campbell Sleep Scale', 'Visual Analog Scala', 'Trait-Trait Anxiety Inventory', 'Postpartum Comfort Scale', 'Bristol Breastfeeding Assessment Tool', 'Uterine Involution Evaluation Form', 'Physiological Parameter Form' will be filled in again. . Participants in the control group will not receive massage and will receive routine nursing care. Pain, sleep, comfort, breastfeeding and heart rate, body temperature, anxiety, uterine involution, oxygen saturation, respiratory rate, blood pressure physiological parameters of women in the control group will be measured at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who gave birth at the age of 18 and over
* The one who is married
* At least primary school graduate
* Giving by cesarean section
* Those who had a cesarean section with regional anesthesia
* Having a single, healthy newborn at full term
* Those who did not experience any problems during pregnancy
* Pain intensity is 40 mm or more according to the Visual Analogue Scale
* Does not react negatively to any attempt at touch, such as massage
* The tissue integrity in the area to be massaged is complete and healthy
* Women who agree to participate in the research will be included in the study

Exclusion Criteria:

* Those who gave birth by cesarean section before the 37th week of pregnancy
* Having diseases such as heart disease, diabetes, hypertension
* Receiving controlled analgesia after cesarean section
* Having received a psychiatric diagnosis such as anxiety and depression
* Those who develop postpartum complications
* Women who want to leave the research at any stage of the research will be excluded from the research

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The gender required to sample women who gave birth by cesarean section must be female.
Enrollment: 78 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | twenty four hours
  It is used for pain assessment in musculoskeletal and other clinical evaluations. VAS is used to convert some values that cannot be measured numerically into numerical values. It is a frequently used measurement tool because it is easy to apply and safe. At the left end of the 10 cm long horizontal line are the words 'I have no pain' and at the right end the words 'I have pain'. The individual is told to mark the point on this horizontal line that best expresses the intensity of pain in his body. The distance of the point marked by the individual to the left end is measured and the pain score is determined. As the VAS value approaches 10, the intensity of the pain increases, and as it approaches 0, the intensity decreases. The lowest score from the scale is 0 and the highest score is 10.

SECONDARY OUTCOMES:
Richard-Campbell Sleep Scale | twenty four hours
  The Richard-Campbell Sleep Scale was developed to evaluate sleep quality, and its Turkish validity and reliability were tested. The scale consists of 6 items that evaluate the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake when waking up, the quality of sleep and the noise level in the environment. The items in the scale are evaluated by scoring between 0-100. Scale scoring is done by dividing the total score from the first five items of the scale by 5. A score between '0-25' from the scale indicates 'very poor sleep', and a score between '76-100' indicates 'very good sleep'. Scale score is directly proportional to sleep quality. Accordingly, as the score increases, sleep quality also increases. Cronbach's alpha coefficient was found to be 0.82 in the original form of the scale and 0.91 in the Turkish form.
Postpartum Comfort Scale | twenty four hours
  Postpartum Comfort Scale is a scale developed in the form of a 5-point Likert to measure comfort level. Scoring and expressions ranging from "completely agree" (5 points) to "strongly disagree" (1 point) were made for all scale items. The expression "I completely agree" expresses the highest comfort (5 points) in positive sentences, and the lowest comfort (1 point) in negative sentences. In this case, the highest score to be obtained from the scale is 170 and the lowest score is 34. The increase in the average score obtained from the scale indicates that the comfort level also increases. Cronbach's Alpha reliability coefficient of the scale is total Postpartum Comfort Scale was found to be 0.78 for.
Bristol Breastfeeding Assessment Tool | twenty four hours
  Bristol Breastfeeding Assessment Scale (BBAT) is used to evaluate the adequacy of breastfeeding in the postpartum period. The scale is observed while the mother is breastfeeding, and the application time is on average 5-10 minutes. The measurement tool is a Likert-type scale consisting of four items: 'positioning', 'holding', 'sucking' and 'swallowing'. In the scoring of the scale, each item is worth 0-2 points. The calculation method is to add up all the scores from the scale items. The lowest score from the scale is 0, the highest score is 8. The scale does not have a cut-off point. A low score indicates that breastfeeding is not effective, and a high score indicates that breastfeeding is effective. There is no need to observe breastfeeding from start to finish to make an evaluation; observation can be made at any time during breastfeeding.
State Anxiety Inventory (STAI Form) | twenty four hours
  The State Anxiety Inventory is a Likert-type four-degree scale ranging from "Not at all" to "Completely". There are two types of statements in the State-Trait Anxiety Inventory. Inverted expressions, those with a weight of 1 turn into 4, and those with a weight of 4 turn into 1. Answers with a value of 4 on 33 direct statements indicate high anxiety. In reversed expressions, answers with a value of 1 indicate high anxiety, and answers with a value of 4 indicate low anxiety. After finding the separate total weights of direct and reverse expressions, the total weight score of reverse expressions is subtracted from the total weight score obtained for direct expressions. This value is 50 for the State Anxiety Inventory and 35 for the Trait Anxiety Inventory. The last value obtained is the individual's anxiety score. The scores obtained from both scales theoretically range between 20 and 80. A large score indicates a high level of anxiety, a small score indicates a low level of anxiety.
Uterine Involution Evaluation Form | twenty four hours
  Immediately after uterine involution and delivery of the placenta, the apex of the fundus is located in the midline, between the symphysis and the umbilicus. 6-12 hours after birth, the fundus is at the umbilicus level and the height of the fundus decreases approximately 1 cm every day. Uterus Involution Evaluation Form is a form prepared by the researcher in line with the literature, in which the measurement of the length of the uterus is recorded and the uterine involution process of postpartum women is evaluated. To evaluate the involution of the uterus, the distance between the fundus of the uterus and the symphysis pubis will be measured with a tape measure. Uterine length will be measured when the women's bladder is empty and the same tape measure will be used in all measurements.
Physiological Parameter Form | twenty four hours
  Physiological parameters are important indicators in the management of the postpartum period and in determining the treatment protocol. Heart rate, body temperature, oxygen saturation, respiratory rate and blood pressure, which are stated as basic life parameters, are parameters that indicate the health status of the person. Although physiological parameter values vary individually, according to the standards determined by the World Health Organization, blood pressure is 8/120 mm/hg, body temperature 36.1°C-37.2°C, pulse rate of 60-100 beats per minute, respiratory rate of 12-20 per minute, and oxygen saturation of 95-100% are considered normal. For this purpose, the Physiological Parameter Form includes heart rate, body temperature, oxygen saturation, respiratory rate and blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Esra GÜLER EG PhD student, Principal Investigator — Ordu University
Locations (1):
- Fatsa State Hospital, Fatsa, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) can be shared with other researchers via e-mail sent to me after the study is completed, when a meta-analysis study will be conducted.